CLINICAL TRIAL: NCT01973699
Title: Surgeon Determined Visualization in Shoulder Arthroscopy: A Randomized, Blinded, Controlled Trial Comparing Irrigation Fluid With and Without Epinephrine
Brief Title: Visualization in Shoulder Arthroscopy With and Without Epinephrine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Luke's Hospital, Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: SLHN 2012-61
Record Dates: First submitted 2013-10-25; First posted 2013-10-31 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Visualization in Shoulder Arthroscopy
Keywords: shoulder arthroscopy, epinephrine, visualization

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- With Epinephrine (Placebo Comparator): Patients undergoing shoulder arthroscopy with epinephrine in their irrigation as standardly performed
  Interventions: Other: visualization in shoulder arthroscopy
- Without Epinephrine (Experimental): Patients undergoing shoulder arthroscopy without epinephrine in their irrigation fluid as typically done
  Interventions: Other: visualization in shoulder arthroscopy

INTERVENTIONS:
Other: visualization in shoulder arthroscopy — Evaluating the effect of performing shoulder arthroscopy with and without epinephrine on visualization

SUMMARY:
Adequate visualization during shoulder arthroscopy is of great importance for the procedure to be efficiently and effectively performed. The use of dilute epinephrine in irrigation fluid has been historically utilized to help with visualization. Given the potential safety issues documented in the literature related to epinephrine use, as well as the significant improvements in technique and instrumentation over the last decade, the need for this additive should be reexamined. The objective of the current study was to compare surgeon determined visualization in shoulder arthroscopy using irrigation fluid with and without epinephrine.

ELIGIBILITY:
Inclusion Criteria:

All patients requiring shoulder arthroscopy

Exclusion Criteria:

none

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2012-11; Primary Completion 2013-04 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Visualization | November 1, 2012- April 1, 2013 (5 months)
  surgeon determined visualization during shoulder arthroscopy as judged by a VAS

SECONDARY OUTCOMES:
Fluid Use | November 1, 2012-April 1, 2013 (5 months)
  fluid used during arthroscopy
Operative time | November 1, 2012-April 1, 2013 (5 months)
  operative time

CONTACTS AND LOCATIONS:
Overall Officials: Gregory F Carolan, MD, Principal Investigator — St. Luke's University Hospital and Health Network
Locations (1):
- St. Luke's University Hospital, Bethlehem, Pennsylvania, United States